CLINICAL TRIAL: NCT07226362
Title: A Phase-1, Open-label Randomized, 4-treatment, 4-period Crossover Study to Evaluate the Pharmacokinetics, Relative Bioavailability, Safety and Tolerability of Single Doses of Dihydroergotamine Mesylate (DHE) Inhalation Powder, DHE Intravenous (IV), and DHE Nasal Spray in Healthy Adult Subjects.
Brief Title: A Study Evaluating the Safety, Tolerability and Pharmacokinetics of ASY202 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aspeya Switzerland SA (Industry)
Responsible Party: Sponsor
Organization: Aspeya, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VFC202-102
Record Dates: First submitted 2025-10-28; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Safety, and Tolerability
Keywords: Dihydroergotamine mesylate; Inhalation powder
MeSH Terms: interventions — Dihydroergotamine; Metoclopramide

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be enrolled and randomized on Day 1 to one of the 4 treatment sequences composed of 4 periods of the crossover design.
Masking Description: None (open-label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: inhaled DHE low dose (Experimental): Low dose of DHE inhalation powder
  Interventions: Combination Product: DHE inhalation powder low dose administered via dry powder inhaler (DPI) device
- Treatment B: inhaled DHE high dose (Experimental): High dose of DHE inhalation powder
  Interventions: Combination Product: DHE inhalation powder high dose administered via dry powder inhaler (DPI) device
- Treatment C: intravenous DHE (Active Comparator): 1 mg DHE injected intravenously
  Interventions: Drug: DHE injected intravenously (1 mg); Drug: Metoclopramide 10mg
- Treatment D: intranasal DHE (Active Comparator): 2 mg DHE nasal spray (Migranal®)
  Interventions: Drug: DHE 2 mg administered by nasal spray (Migranal®)

INTERVENTIONS:
Combination Product: DHE inhalation powder low dose administered via dry powder inhaler (DPI) device — The DHE inhalation powder is a pre-metered drug-device combination product containing DHE dry powder low dose formulation for oral inhalation
  Arms: Treatment A: inhaled DHE low dose
Combination Product: DHE inhalation powder high dose administered via dry powder inhaler (DPI) device — The DHE inhalation powder is a pre-metered drug-device combination product containing DHE dry powder high dose formulation for oral inhalation
  Arms: Treatment B: inhaled DHE high dose
Drug: DHE injected intravenously (1 mg) — A single dose of DHE injection consists of 1 mg/mL ampoule of DHE solution for slow intravenous administration.
  Arms: Treatment C: intravenous DHE
Drug: DHE 2 mg administered by nasal spray (Migranal®) — A single vial of DHE nasal spray (Migranal®) contains 1 mL of 4 mg/mL DHE solution.
  Arms: Treatment D: intranasal DHE
Drug: Metoclopramide 10mg — To prevent nausea caused by IV administration of DHE, participants will receive antiemetic pre-medication with metoclopramide 10 mg administered by slow intravenous push over 1-2 min, given 5 to 10 minutes prior to IV DHE dosing.
  Arms: Treatment C: intravenous DHE

SUMMARY:
A Phase 1 clinical trial to evaluate the pharmacokinetics, relative bioavailability, safety and tolerability of DHE inhalation powder delivered by dry powder inhaler, DHE IV, and DHE nasal spray.

DETAILED DESCRIPTION:
This is an open-label, randomized, 4-treatment, 4-period crossover study to evaluate the PK, relative BA, safety, and tolerability of single doses of study medication in healthy adult subjects.

Following screening, eligible subjects will be enrolled and randomized to one of the 4 treatment sequences. Subjects will receive single doses of DHE inhalation powder (low dose and high dose), DHE IV (1 mg) and DHE nasal spray (2 mg).

Subjects will be administered one treatment in each period according to their assigned sequence. Each subject will receive all 4 treatments in the study.

During each treatment period subjects will remain in the clinical research unit for 3 days, until completion of the 48-hour post-dose assessments.

Subjects will return for their next treatment period after at least 7 days washout after the administration of their previous treatment until all periods have been completed in their sequence.

A follow-up will be conducted on Day 7 after the last dose in the study to assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following criteria to be included in the study:

  1. Male or female, ≥ 18 and ≤ 55 years of age, with body mass index (BMI) >18.5 and < 32.0 kg/m2
  2. Healthy subjects
  3. Female subjects of non-childbearing potential or childbearing potential willing to use protocol required methods of contraception
  4. Current non-smoker
  5. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  1. Positive pregnancy test or lactating female subjects at screening or on Day 1 of each treatment period
  2. Clinically significant abnormal laboratory or serology test results
  3. History or current diagnosis of uncontrolled or significant cardiac disease
  4. Significant risk factors for cardiovascular disease
  5. Subject with abnormal lung function at screening
  6. History or current diagnosis of lung disease e.g. asthma, COPD
  7. Known allergic reactions, hypersensitivity or contraindications to DHE, other ergot-derived products or to any excipient
  8. History of drug or alcohol abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the curve (AUC 0-t) of DHE | For each of the 4 treatment periods on baseline and post-dose measurements from 2 min up to 48 hrs
  Area under the concentration-time curve from time zero until the last observed plasma concentration of DHE (AUC 0-t)
Pharmacokinetics: Area under the curve (AUC 0-inf) of DHE | For each of the 4 treatment periods on baseline and post-dose measurements from 2 min up to 48 hrs
  Area under the concentration-time curve from time zero to infinity (extrapolated) of plasma concentrations of DHE (AUC 0-inf)
Pharmacokinetics: Peak plasma concentration (C max) of DHE | For each of the 4 treatment periods on baseline and post-dose measurements from 2 min up to 48 hrs
  Maximal observed plasma concentration of DHE (C max)

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the curve (AUC 0-t) of 8'-OH-DHE | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Area under the concentration-time curve from time zero until the last observed plasma concentration of 8'-OH-DHE (AUC 0-t)
Pharmacokinetics: Area under the curve (AUC 0-inf) of 8'-OH-DHE | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Area under the concentration-time curve from time zero to infinity (extrapolated) of plasma concentrations of 8'-OH-DHE (AUC 0-inf)
Pharmacokinetics: Peak plasma concentration (C max) of 8'-OH-DHE | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Maximal plasma observed concentration of 8'-OH-DHE (C max)
Pharmacokinetics: Time of peak maximal concentration (T max) of DHE and 8'-OH-DHE | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Time when the maximal plasma concentration of DHE and 8'-OH-DHE are observed (T max)
Pharmacokinetics: Terminal elimination half-life (T 1/2 el) of DHE and 8'-OH-DHE | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Terminal elimination half-life of plasma concentrations of DHE and 8'-OH-DHE (T 1/2 el)
Pharmacokinetics: Area under the curve (AUC 0-30 min) of DHE | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Area under the concentration-time curve from time zero to 30 min of plasma concentrations of DHE (AUC 0-30min)
Pharmacokinetics: Area under the curve (AUC 0-2 hours) of DHE | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Area under the concentration-time curve from time zero to 2 hours of plasma concentrations of DHE (AUC 0-2 hours)
Pharmacokinetics: Apparent clearance of DHE (CL/F) | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Apparent clearance of DHE (CL/F) for DHE inhalation powder and DHE nasal spray Migranal®
Pharmacokinetics: Clearance of DHE (CL) | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Clearance of DHE for intravenous DHE (CL)
Pharmacokinetics: Apparent volume of distribution of DHE (Vz/F) | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Apparent volume of distribution (Vz/F) during terminal phase of DHE for DHE inhalation powder and DHE nasal spray Migranal®
Pharmacokinetics: Volume of distribution of DHE (Vz) | For each of the 4 treatment periods on Baseline and post-dose measurements from 2 min up to 48 hrs
  Volume of distribution (Vz) of DHE intravenous
Safety: Number of participants with adverse events | From the time of signing the informed consent until the last visit on Day 7 after the last treatment period
  Adverse events will be recorded and evaluated for their seriousness, severity and relationship to the study drug
Safety: Blood pressure in mmHg | Baseline and post-dose measurements from 10 min up to 48 hrs for each of the 4 treatment periods
  The changes from baseline in systolic and diastolic blood pressure will be assessed
Safety: Heart rate in beats/min | Baseline and post-dose measurements from 10 min up to 48 hrs for each of the 4 treatment periods
  The changes from baseline in heart rate will be assessed
Safety: Respiratory rate in breaths/min | Baseline and post-dose measurements from 10 min up to 48 hrs for each of the 4 treatment periods
  The changes from baseline in respiratory rate will be assessed
Safety: Oral body temperature in degree Celsius | Baseline and post-dose measurements from 10 min up to 48 hrs for each of the 4 treatment periods
  The changes from baseline in oral body temperature will be assessed
ECG PR interval in msec | Baseline and post-dose measurements from 10 min up to 4 hrs for each of the 4 treatment periods
  The changes from baseline in 12-lead ECG PR interval will be assessed
ECG QRS complex in msec | Baseline and post-dose measurements from 10 min up to 4 hrs for each of the 4 treatment periods
  The changes from baseline in 12-lead ECG QRS complex will be assessed
ECG QT interval in msec | Baseline and post-dose measurements from 10 min up to 4 hrs for each of the 4 treatment periods
  The changes from baseline in 12-lead ECG QT interval and Fridericia's corrected QT interval will be assessed
Physical examination | At screening, and for each of the 4 treatment periods at baseline, and post-dose at day 2 and day 3
  Physical examination (including oral cavity, nasal cavity and injection site examination) will be performed
Lung function by spirometry : Forced Expiratory Volume in 1 sec in % of predicted normal (FEV1 ) | At screening, and for each of the 4 treatment periods at pre-dose, and post-dose up to 48 hours
  Effect of DHE on lung function will be measured by collecting FEV 1 pre- and post-dose at specified timepoints and will be analyzed by FEV1 < 70 % of predicted normal and/or comparison of pre- and post-dose > 20 % decline in FEV1.
Lung function by spirometry : Forced Vital Capacity (FVC) in liters | At screening, and for each of the 4 treatment periods at pre-dose, and post-dose up to 48 hours
  Effect of DHE on lung function will be measured by collecting Forced Vital Capacity pre- and post-dose at specified timepoints
Lung function by spirometry : FEV1/FVC ratio | At screening, and for each of the 4 treatment periods at pre-dose, and post-dose up to 48 hours
  Effect of DHE on lung function will be measured by collecting the FEV1/FVC ratio pre- and post-dose at specified timepoints
Lung function by spirometry : Forced Expiratory Flow 25-75 in % | At screening, and for each of the 4 treatment periods at pre-dose, and post-dose up to 48 hours
  Effect of DHE on lung function will be measured by collecting the mean Forced expiratory Flow between 25% and 75% of the forced vital capacity pre- and post-dose at specified timepoints
Clinical laboratory tests blood and urine | At screening, and for each of the 4 treatment periods at pre-dose, and post-dose up to 48 hours
  Change from baseline in clinical laboratory tests (including hematology, biochemistry, coagulation, and urinalysis) will be analyzed at different timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Alliance for Multispecialty research (AMR), Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No